CLINICAL TRIAL: NCT03888248
Title: Whole-body Vibration Training Compared to Muscle-strengthening Exercises Alone in Improving Muscle Function in Children With Neurofibromatosis Type 1
Brief Title: Whole-body Vibration in Children With Neurofibromatosis Type 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: Manchester Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B00472
Record Dates: First submitted 2019-03-20; First posted 2019-03-25 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Neurofibromatosis Type 1; Muscle Weakness
Keywords: Neurofibromatosis Type 1; Whole-body vibration; Muscle weakness
MeSH Terms: conditions — Neurofibromatosis 1; Muscle Weakness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercises (Active Comparator): Daily muscle-strengthening exercises
  Interventions: Other: Muscle strengthening exercises
- Whole-body vibration + exercises (Experimental): Home-based whole-body vibration therapy plus daily muscle-strengthening exercises
  Interventions: Device: Whole-body vibration; Other: Muscle strengthening exercises

INTERVENTIONS:
Device: Whole-body vibration — Home-based whole-body vibration therapy by standing on Galileo Med 15 platform for 9 mins twice a day for 5 days per week
  Arms: Whole-body vibration + exercises
Other: Muscle strengthening exercises — Daily muscle strengthening exercises to be performed at home following a group education session by paediatric physiotherapist

SUMMARY:
It is known that children with NF1 can have weak muscles and suffer from tiredness. It is also known that in similar conditions affecting children's muscles, standing on a vibration device for a few minutes each day can strengthen muscles and improve their ability to perform day-to-day activities. The investigators believe this vibrating platform can be used to strengthen the muscles of children with NF1 also, beyond standard exercises, and therefore allow them to perform day-to-day activities better, do more activity and feel less tired.

If families are keen to take part in this study, the investigators will first need to check they are suitable for the trial. This will be based on the participant's age (6-16 years), their other medical problems that would affect use of the vibration device or tests to assess how effective it is, and their level of muscle weakness.

Once families have agreed to take part, participants will be randomised either to receive a muscle-strengthening exercise session delivered by a physiotherapist that children with weak muscles should continue to perform daily for the next 6 months; or to receive a vibration device to take home and use for a few minutes 5 days a week for 6 months as well as the exercises.

All participants will be invited to attend for a variety of activities and tests, just before starting the trial and 6 months later at the end of the trial to see if there is any benefit from the vibration device. The investigators will repeat these tests again 3 months later, to see if any benefits observed remain, even after the device is removed. They will involve jumping, hopping and balancing on a board, gripping a machine as hard and as long as possible, being fitted with a device that measures activity for 7 days, walking as far as possible for 6 minutes, scanning muscles using MRI, completing a tiredness and general well-being questionnaires, and parents completing a questionnaire of the participant's attention and intellect. The jumping will also be performed 3 months into the study, to see if there is any early improvement in this key test.

All participants will be given full details of what the trial involves before taking part. As with any other trial, participants and their families are free to stop taking part at any time. Although the investigators do not anticipate any safety issues, if any do arise, the families will be asked to contact the trial team.

DETAILED DESCRIPTION:
Children with neurofibromatosis type 1 (NF1) have been shown in many studies to have reduced muscle mass, strength and function. This could potentially contribute to the fatigue and low quality of life reported in these children. However, to date interventions to improve muscle mass, strength and function in these children have not been established. Whole body vibration (WBV) has been demonstrated to improve walking speed and distance, muscle mass and strength, spasticity and balance in children with other neuromuscular conditions.

In this proposed preliminary matched-pairs interventional trial, the investigators aim to identify whether a home-based WBV therapy programme (9 minutes twice daily for 5 days per week) in addition to standard daily muscle-strengthening exercises improves muscle mass, strength and function over a six month period in children with NF1 aged 6-16 years, compared to daily muscle-strengthening exercises alone. Participants must have evidence of poor muscle strength, with grip force used to assess for this. Key exclusion criteria include significant learning difficulty or autistic spectrum disorder which would create difficulty in use of the WBV device, focal skeletal abnormalities and contraindications to WBV therapy.

The primary outcome measure will be dynamic muscle function using mechanography to measure peak power per kilogram on single two-legged jump.

Secondary/exploratory outcome measures include the 6-minute walk test (to assess lower limb muscle function and mobility), accelerometer data (as a surrogate marker of type and duration of physical activity), hand-held dynamometry (to assess upper limb grip force and endurance), measures on mechanography other than jumping power (to further assess dynamic muscle function), MRI for muscle cross-sectional area and signal intensity, fatigue and general well-being questionnaires and parental reports of attention and cognition.

These measures will be undertaken at baseline, on completion of intervention at 6 months, and again 3 months after to identify whether there is any sustained effect of the intervention following removal. Halfway through the intervention period (3 months), participants will also be invited just to complete the primary outcome of single two-legged jump on ground reaction force plate, as an interim measure.

The investigators hypothesise that WBV therapy will result in increased muscle mass and passive muscle strengthening of the lower limbs, which will translate into better muscle function in the lower limbs compared to baseline data and control group. As it is hypothesised that muscle weakness contributes to the fatigue demonstrated in children with NF1, the investigators would expect to see an improvement in their fatigue scores, which, combined with greater muscle strength, will translate into greater physical activity. The investigators hypothesise that WBV may also have an impact on muscle function in the upper limbs through central sensory stimulation and neuronal rewiring. Many children with NF1 have evidence of attention problems, and the investigators hypothesise that this may improve with WBV, again through central neuronal rewiring.

The trial will be conducted in compliance with this protocol, Good Clinical Practice (GCP) and applicable regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Neurofibromatosis Type 1 (confirmed by NIH consensus criteria)
* Grip force less than -1 SDS according to age- and gender-matched normative data

Exclusion Criteria:

* Focal skeletal abnormalities (pseudoarthrosis, kyphoscoliosis likely to require surgery, known spondylolisthesis)
* Significant autistic spectrum disorder or learning difficulties (neurodevelopmental age less than 6 years)
* Inability to adequately weight-bear or balance on vibrating platform
* Lower limb plexiform causing limb length discrepancy
* Contraindications to use of whole-body vibration device (acute thrombosis, implants in activated regions of the body, acute inflammation of the locomotor system, herniae, propensity to fragility fractures or fracture within the past 3 months, history of renal calculi, epilepsy)

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Change in peak power per kilogram on single two-legged jump using Leonardo Mechanography Ground Reaction Force Plate | Baseline, 6 months
  Change from baseline to 6 months of peak power per kilogram of single two-legged jump using Leonardo Mechanography Ground Reaction Force Plate. Power will be measured in watts.

SECONDARY OUTCOMES:
6 minute walk test | Baseline, 6 months, 9 months
  Distance in metres walked during 6 minutes
Accelerometer (duration) | Baseline, 6 months, 9 months
  Duration of activity in minutes over 7 days using accelerometer
Accelerometer (intensity) | Baseline, 6 months, 9 months
  Intensity of activity (accelerometer counts per minute) over 7 days using accelerometer
PedsQL Multi-dimensional Fatigue Scale | Baseline, 6 months, 9 months
  Total score from age-appropriate validated questionnaire that asks for perceived fatigue within the domains of 'General', 'Sleep/Rest' and 'Cognitive'. Each domain consists of 6 questions, with participants/parents rating each question from 0 to 4 (therefore total score can range from 0 to 72). A higher total score indicates greater fatigue (i.e. worse outcome)

OTHER OUTCOMES:
Peak force (newtons) per kilogram on multiple one-legged hop using Leonardo Mechanography Ground Reaction Force Plate | Baseline, 6 months, 9 months
Efficiency of single two-legged jump using Leonardo Mechanography Ground Reaction Force Plate | Baseline, 6 months, 9 months
  Efficiency is calculated by the Leonardo software by comparing peak force and peak power, and is an indicator of movement velocity and co-ordination. The software will automatically calculate z-score (based on weight, age and gender), which will be used for analysis
Balance tasks | Baseline, 6 months, 9 months
  Most complex balance task that can be performed for 10 seconds will be recorded (increasing in complexity from Romberg stance, to semi-tandem stance, to tandem stance, to balancing on one foot). This will be performed on Leonardo Mechanography Ground Reaction Force Plate
Path length using Leonardo Mechanography Ground Reaction Force Plate | Baseline, 6 months, 9 months
  Path length in centimetres of the completed balance tasks
Ellipse area using Leonardo Mechanography Ground Reaction Force Plate | Baseline, 6 months, 9 months
  Ellipse area in centimetres squared of the completed tasks
Maximal hand grip force | Baseline, 6 months, 9 months
  Maximal hand grip force (newtons) using hand-held dynamometry
Sustained grip force | Baseline, 6 months, 9 months
  Sustained grip force (newtons) over 10 seconds using hand-held dynamometry
Magnetic resonance imaging of right calf muscle | Baseline, 6 months, 9 months
  Cross-sectional area in centimetres squared of calf muscles in right leg
Magnetic resonance imaging of right mid-thigh muscle | Baseline, 6 months, 9 months
  Cross-sectional area in centimetres squared of mid-thigh muscles in right leg
Magnetic resonance imaging - signal intensity | Baseline, 6 months, 9 months
  Average signal intensity of right leg muscle on MRI
Child Outcome Rating Scale | Baseline, 6 months, 9 months
  Total score from non-validated visual analog scale of participant's perception of lifestyle and well-being. This will assess participant's perception of 6 domains: 'Mood and emotional well-being', 'Tiredness/fatigue', 'Hobbies/interests/activities', 'School', 'Attention/concentration' and ''Overall'. Each domain is on a 10cm rule, therefore total score can range from 0 to 60. A higher score indicates better well-being (i.e. better outcome).
Conners Parent Rating Scale | Baseline, 6 months, 9 months
  Total score on validated questionnaire for parental report of attention deficit hyperactivity disorder (ADHD) symptomatology, within domains of 'Inattention', 'Hyperactivity/impulsivity', 'Learning problems', 'Executive functioning', 'Aggression' and 'Peer relations'. There are 45 questions, each rated on a scale of 0 to 3 (therefore total score can range from 0 to 135). A higher score indicates greater features of ADHD (i.e. worse outcome).
Persistence of changes in primary outcome on withdrawal of intervention | Baseline, 9 months
  Change from baseline to 9 months (i.e. 3 months after withdrawal of intervention) of peak power (in watts) per kilogram of single two-legged jump using Leonardo Mechanography Ground Reaction Force Plate
Evidence of early changes in primary outcome | Baseline, 3 months
  Change from baseline to 3 months (i.e. half way through intervention) of peak power (in watts) per kilogram of single two-legged jump using Leonardo Mechanography Ground Reaction Force Plate

CONTACTS AND LOCATIONS:
Overall Officials: Zulf Mughal, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- Manchester University Hospitals NHS Foundation Trust, Manchester, United Kingdom